CLINICAL TRIAL: NCT07104019
Title: Evaluation of the Effectiveness of Blood Concentrate Biofiller in Thickening the Gingival Phenotype Around Natural Teeth
Brief Title: Biofiller and Gingival Phenotype Thickening
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Kubra Aral, Associate Professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-3647
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Gingival Recession; Gingival Diseases; Gingival Inflammation
Keywords: biofiller; gingival phenotype modification; connective tissue graft
MeSH Terms: conditions — Gingival Recession; Gingival Diseases; Gingivitis

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, controlled, parallel-arm clinical trial designed to compare the efficacy of biofiller (albumin-enriched PRF) injection and connective tissue grafting in increasing gingival thickness in patients with thin periodontal phenotype.
Who Masked: Outcomes Assessor
Masking Description: While the study is open-label for participants and care providers due to the nature of the interventions, clinical measurements and soft tissue scans will be evaluated by a blinded assessor who is unaware of the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofiller Injection Group (Experimental): Patients in this group will receive biofiller composed of albumin-enriched platelet-poor plasma (PPP) and concentrated platelet-rich fibrin (c-PRF), prepared from the patient's autologous blood. After a tunneling procedure in the mandibular anterior region (canine-to-canine), 0.5 mL of biofiller will be injected per tooth
  Interventions: Procedure: Biofiller Injection
- connective tissue graft group (Active Comparator): Participants in this group will undergo a minimally invasive tunneling surgical procedure in the mandibular anterior region (canine to canine). Autogenous connective tissue grafts (CTG) will be harvested from the patient's palate and placed under the gingiva through the tunnel to increase gingival thickness. The graft will be stabilized without vertical releasing incisions. No biomaterials or adjunctive agents will be used. All procedures will be performed under local anesthesia by an experienced periodontist.
  Interventions: Procedure: connective tissue graft

INTERVENTIONS:
Procedure: Biofiller Injection — Biofiller will be prepared by heating the platelet-poor plasma (PPP) component obtained from peripheral blood, which is then mixed with concentrated PRF (c-PRF). After creating a surgical tunnel in the mandibular anterior region (canine to canine), 0.5 mL of the prepared biofiller will be injected into each tooth region under the gingiva. The procedure is performed under local anesthesia and aims to increase gingival thickness in patients with a thin periodontal phenotype.
  Other Names: Albumin-enriched Platelet-Rich Fibrin injection
  Arms: Biofiller Injection Group
Procedure: connective tissue graft — A connective tissue graft will be harvested from the palatal donor site and placed under the gingiva using a minimally invasive tunneling technique in the mandibular anterior region (canine to canine). The procedure will be performed under local anesthesia and aims to increase gingival thickness. No biomaterials or adjunctive agents will be used.
  Other Names: Autogenous Connective Tissue Graft
  Arms: connective tissue graft group

SUMMARY:
The periodontal phenotype is defined as the combination of the gingival phenotype and the thickness of the buccal bone plate (bone morphotype). The gingival phenotype refers to the gingival thickness (GT) and the width of the keratinized tissue (KTW). A gingival thickness of ≤1 mm is classified as a thin phenotype, whereas a thickness >1 mm is considered a thick phenotype. Thin gingival biotypes tend to show more pronounced responses to inflammation, restorations, trauma, and parafunctional habits. Various methods are used to assess gingival thickness, including transgingival probing (TP), ultrasonic measurements, cone-beam computed tomography (CBCT) scans, visual assessment, and colored biotype probes (CBP). Periodontal plastic procedures performed using autogenous grafts such as connective tissue grafts (CTG) and free gingival grafts (FGG), or biomaterials such as acellular dermal matrices (ADM) and collagen matrices (CM), are known to significantly increase GT and the amount of keratinized tissue. However, creating a second surgical site in the oral cavity during these procedures may compromise patient comfort, prompting researchers to explore alternative methods. Additionally, the effectiveness of synthetic biomaterials has been found to be lower than that of autogenous grafts.

Platelet-rich concentrates have been used as a minimally invasive procedure for the past thirty years, showing a high capacity to release growth factors that support tissue regeneration. While platelet-rich plasma (PRP), as the first-generation platelet concentrate, is widely used, platelet-rich fibrin (PRF) has been increasingly applied across various fields of medicine and dentistry due to its ability to release more growth factors over a longer period, resulting in better clinical outcomes. PRF is a highly biocompatible material composed of autologous cells and growth factors entrapped in a fibrin matrix, and has been shown to degrade more slowly over time compared to conventional PRP. One of the main reported disadvantages of PRF (and especially PRP) is its relatively rapid resorption, typically within 2-3 weeks. Biofiller is an autologous material derived from the patient's own blood and includes platelet-poor plasma (PPP) and concentrated platelet-rich fibrin (PRF). The PPP component is heated to become enriched with albumin, thereby prolonging its resorption time. The PRF portion contains autologous cells and growth factors. However, conventional PRF is typically resorbed within 2-3 weeks, limiting its clinical application. Recent studies have shown that the resorption time of biofiller-a combination of PPP and PRF-can exceed 4 months.

The aim of this study is to compare the effectiveness of biofiller with connective tissue graft in increasing gingival thickness in patients with a thin gingival phenotype. A total of 34 patients (17 patients in each group) will be enrolled. Tunnel surgery will be performed to all participants and test group will receive biofiller only once. Control group will receive connective tissue surgery. Clinical parameters obtained from our patients at baseline and at follow-up visits at 1, 3, and 6 months - including gingival thickness (GT), keratinized tissue width (KTW), and soft tissue measurements assessed via intraoral scanners - will be compared.

DETAILED DESCRIPTION:
The periodontal phenotype is determined by gingival thickness (GT), the width of keratinized tissue (KTW), and buccal bone thickness. A thin phenotype (GT ≤1 mm) is more susceptible to inflammation, trauma, and surgical complications. To increase soft tissue thickness, autogenous grafts such as connective tissue grafts (CTG) or biomaterials like collagen matrices are used. However, autogenous grafts require a second surgical site, which may reduce patient comfort.

Biofiller is a novel autologous material prepared by heating platelet-poor plasma (PPP) and combining it with concentrated platelet-rich fibrin (c-PRF), resulting in a biocompatible gel with prolonged resorption time and regenerative potential.

This randomized controlled clinical trial aims to compare the effectiveness of Biofiller versus connective tissue graft in increasing gingival thickness in patients with a thin gingival phenotype.

In the literature, several clinical indications have been proposed for phenotype modification in individuals with a thin phenotype, such as prior to orthodontic treatment, when implant placement is planned, or when a restoration is intended to be placed subgingivally. Therefore, all participants in this study will undergo an orthodontic evaluation prior to treatment.

A total of 34 systemically healthy patients with a thin phenotype in the mandibular anterior region will be enrolled. All participants will undergo a standardized tunneling procedure (canine to canine). The test group will receive a single injection of 0.5 mL Biofiller per tooth, while the control group will receive a connective tissue graft.

To ensure standardization, individuals with Class II or Class III orthodontic anomalies will be excluded. Lateral cephalometric radiographs will be obtained to measure buccal bone thickness at three points per tooth, and an average value will be calculated. Only patients with a Class I skeletal relationship and an orthodontic treatment indication will be included.

Clinical parameters including GT, KTW, and digital soft tissue thickness (via intraoral scanner) will be recorded at baseline, and at 1, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years
* Systemically healthy individuals
* Presence of thin gingival phenotype in the mandibular anterior region (canine to canine)
* No medications that affect wound healing
* No history of bleeding disorders
* No known allergy to anti-inflammatory drugs
* Not pregnant or breastfeeding
* Willingness to participate and provide informed consent
* Non-smoker

Exclusion Criteria:

* Systemic diseases (e.g., diabetes, hypertension, cancer, etc.)
* Use of medications that may affect healing (e.g., corticosteroids, immunosuppressants)
* History of radiotherapy or chemotherapy
* Pregnancy or breastfeeding
* Poor oral hygiene
* Refusal to participate
* Age under 18 years
* Smoking
* Presence of Class II or Class III orthodontic anomalies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2025-11-03 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Gingival Thickness (GT) | Baseline, 1 month, 3 months, 6 months
  Gingival thickness will be measured in the mandibular anterior region (canine to canine) using a digital caliper and intraoral scanner. The change in GT from baseline to each follow-up visit will be assessed to evaluate the efficacy of biofiller versus connective tissue graft in augmenting gingival thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Kubra Aral, PhD, Principal Investigator — Inonu University
Locations (1):
- Inonu university, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be made available to other researchers due to ethical and privacy considerations.